CLINICAL TRIAL: NCT03726281
Title: Phase II Multi-institutional Proof of Concept Single-arm Trial of Nivolumab in the Treatment of Patients With Platinum Recurrent or Refractory Metastatic Germ Cell Tumors
Brief Title: Nivolumab in Platinum Recurrent or Refractory Metastatic Germ Cell Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: End of Agreement between BMS and SGHL
Sponsor: Hospital Beatriz Ângelo (Other)
Collaborators: Universidade Nova de Lisboa (Other); Bristol-Myers Squibb (Industry); Instituto de Patologia e Imunologia Molecular da Universidade do Porto (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBA_001
Record Dates: First submitted 2018-10-11; First posted 2018-10-31 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Germ Cell Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- single-arm trial of Nivolumab (Experimental): Multi-institutional, single arm phase II trial with Simon's optimal two-stage design, to evaluate the clinical benefit of Nivolumab monotherapy in patients with platinum-recurrent or platinum-refractory metastatic GCT. No randomization or blinding is involved.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg, IV

SUMMARY:
To assess the clinical activity of nivolumab monotherapy, as measured by the investigator-assessed clinical benefit rate (CBR), in patients with platinum-recurrent or platinum-refractory metastatic germ cell tumors (GCT). CBR is defined by sum of complete responses (CR), partial responses (PR) and stable disease (SD) for at least 3 months, with stable or declining tumor markers (αFP and HCG), using Response Evaluation Criteria In Solid Tumors (RECIST 1.1).

DETAILED DESCRIPTION:
For patients with testicular GCT, there is no consensus on the most effective treatment for men who relapse after first-line chemotherapy for advanced disease, between salvage conventional cisplatin-based dose chemotherapy and high-dose chemotherapy (HDCT) with autologous hematopoietic stem cell rescue (ASCT). A significant number of patients with recurrent metastatic testicular GCT can still be cured with salvage chemotherapy but long term survival becomes negligible for cisplatin-refractory disease or for patients beyond second relapse. HDCT with ASCT should be considered for patients with recurrent metastatic disease, at least beyond second relapse, although its therapeutic impact has not yet been proven in randomized controlled trials. In contrast, patients with platinum-refractory metastatic GCT and those with recurrent primary mediastinal nonseminomatous GCT (PMNSGCT) are rarely cured by conventional dose salvage chemotherapy.

Immunotherapy with anti-PD-1 and anti-PD-L1 antibodies have demonstrated clinical activity in multiple malignancies, with durable remissions and long-term survivors in patients with metastatic malignant melanoma, non-small cell lung cancer and renal cell cancer, and are being studied in several other tumor types. In GCT a recent study identified PD-L1 expression in 73% of all seminomas and in 64% of all non-seminomas. Patients with low PD-L1 expression had significantly better progression-free survival (PFS) and OS compared to patients with high PD-L1 expression. Frequent expression of PD-L1 in testicular GCT suggests that these patients may benefit from checkpoint inhibitor treatment with anti-PD-1 or anti-PD-L1 antibodies. So far there are only case reports of nine patients with GCT treated with immune check-point inhibitors. One patient, initially diagnosed with metastatic melanoma but subsequently reclassified as non-seminomatous GCT, was treated with a single dose of nivolumab and experienced clinical resolution of lymphadenopathy, decrease in serum tumor markers and a 47% tumor burden reduction by immune-related response criteria. Another report includes seven patients treated with checkpoint inhibitors (nivolumab or pembrolizumab) as a compassionate use off-label treatment attempt for highly-pretreated GCT. Four patients died shortly after beginning treatment due to tumour progression, the remaining three patients received treatment for at least 6 months and long-term tumor response was achieved in two of the three, both of them with tumors highly positive for PD-L1 staining. Another case report was published of a man with a poor-risk nonseminomatous GCT who had disease progression after HDTC/ASCT and had a durable response to immune checkpoint inhibitor.

Recently a single arm phase II trial of pembrolizumab in patients with incurable platinum refractory GCT was presented at ASCO Annual Meeting 2017. This was the first reported trial evaluating immune checkpoint inhibitors in GCT, enrolling 12 male patients age ≥ 18 with metastatic GCT that had progressed after first line cisplatin-based chemotherapy and after at least 1 salvage regimen (CDCT or HDCT). All patients had non-seminoma, the primary tumor site was testis in 11 patients and mediastinum in 1 patient. 5 patients had late relapse (> 2 years) and 6 patients had received prior HDCT. No partial or complete responses were observed, 2 patients achieved radiographic stable disease for 12 and 9 weeks but with continuing rise of AFP, suggesting that Pembrolizumab has no clinically meaningful activity in refractory GCT.

Thus, with limited and conflicting data, further studies with immune checkpoint inhibitors in patients with recurrent metastatic GCT are required.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Male or female, aged 18 years
* Metastatic GCT, seminoma or non-seminoma, previously treated with standard doublet or triplet cisplatin-containing chemotherapy for metastatic disease in: a) second or further relapse from primary testicular, retroperitoneal or ovarian GCT; b) first or further relapse of PMNSGCT; c) primary-refractory GCT (defined as progression within 8 weeks of finishing first-line chemotherapy for advanced GCT); or d) "late relapse" (> 2 years after cisplatinum-containing chemotherapy for metastatic GCT) that is not amenable to surgical resection.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2.
* Evidence of recurrent disease by imaging (CT or MR) or rising tumor markers (αFP or HCG). NOTE: If a rising tumor marker is the only evidence of progressive disease, at least 2 consecutive rising values at least one week apart are needed and alternative causes of increased serum levels of these markers must be excluded (cross reaction with luteinizing hormone (LH) (that can be tested if needed by testosterone suppression of LH), liver disease, use of marijuana, or second primary tumor)
* Received initial cisplatin based combination therapy, such as BEP, EP, VIP, or similar regimens AND, for primary testicular or ovarian GCT, progression after at least one 'salvage' chemotherapy regimen (such as, TIP, VeIP, VIP or high dose chemotherapy with ASCT).
* "Failure" of prior therapy is defined as: a >20% increase in the sum of the longest diameter of target lesions during prior therapy which is not amenable to surgical resection; the presence of new tumor lesions that are not amenable to surgical resection; an increase in αFP or HCG (two separate determinations at least one week apart are required if rising tumor markers are the only evidence of treatment failure) in patients with metastatic disease. NOTE: Patients with clinically growing "teratoma" (normal or declining tumor markers and radiographic progression) should be considered for surgery.
* Use an adequate method of contraception starting with the first dose of study therapy through 5 months after the last dose of study therapy.
* Measurable disease according to RECIST v1.1 obtained by imaging within 28 days prior to registration.
* Non-measurable but evaluable disease associated increasing tumor markers (αFP and HCG) may be eligible, upon review by two PIs.

Exclusion Criteria:

* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* History of allergy or hypersensitivity to study drug components.
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the patient to receive protocol therapy, or interfere with the interpretation of study results.
* Patients with an active, known or suspected autoimmune disease.
* Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Diagnosis of immunodeficiency or current treatment with systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Known history of active Tuberculosis, Human Immunodeficiency Virus (HIV) or active Hepatitis B (i.e. HBsAg reactive) or Hepatitis C (i.e. HCV RNA [qualitative] is detected).
* Treatment with a live vaccine within 30 days of planned start of study therapy. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (i.e. Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Treatment with chemotherapy, targeted small molecule therapy or radiation therapy within 3 weeks prior to study Day 1 or without recovery (ie. ≤ Grade 1) from AEs from such previously administered agents. Patients with alopecia and ≤ Grade 2 neuropathy are an exception to this criterion and qualify for the study.
* Patients with recent major surgery in the previous 14 days prior to starting therapy must have recovered adequately from the toxicity and/or complications from the intervention.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis, other than previously treated brain metastases who are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment) and must be either off corticosteroids or on a stable or decrease dose ≤10 mg daily prednisone (or equivalent).
* Presence of interstitial lung disease or history of pneumonitis requiring treatment with corticosteroids.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR, %) | 3 months
  number of patients with confirmed responses of a. complete responses (CR), disappearance of all imagiologic evidence of disease AND normalization of GCT tumor markers (αFP and HCG), or b. partial responses (PR) and stable diseases (SD) for at least 3 months, with stable, declining or normalized GCT tumor markers (αFP and HCG), divided by the total number of evaluable patients. Tumor response status will be assessed using RECIST 1.1.

SECONDARY OUTCOMES:
CR + marker-negative PR (%) | 3 months
  number of patients with confirmed responses of a. complete responses (CR), disappearance of all imagiologic evidence of disease AND normalization of GCT tumor markers (αFP and HCG), or b. partial responses (PR) and stable diseases (SD) for at least 3 months, with stable, declining or normalized GCT tumor markers (αFP and HCG), divided by the total number of evaluable patients. Tumor response status will be assessed using RECIST 1.1.
CR + PR with stable or declining tumor markers (αFP and HCG) | 3 months
  number of patients with confirmed responses of a. complete responses (CR), disappearance of all imagiologic evidence of disease AND normalization of GCT tumor markers (αFP and HCG), or b. partial responses (PR) and stable diseases (SD) for at least 3 months, with stable, declining or normalized GCT tumor markers (αFP and HCG), divided by the total number of evaluable patients. Tumor response status will be assessed using RECIST 1.1.
Time to response | 6 months
  Median time (measured in months) to achieve a complete response, partial response or stable disease with stable, declining or normalized GCT tumor markers (αFP and HCG)
Duration of clinical response | 24 months
  Median time (measured in months) since complete or partial response or stable disease with stable, declining or normalized GCT tumor markers (αFP and HCG) until progression
Progression Free Survival (PFS) | 24 months
  Median survival time (measured in months) since the first administration of investigational drug until progression of the disease using RECIST 1.1.
Overall Survival (OS) | 24 months
  Median survival time (measured in months) since the first administration of investigational drug until death.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Beatriz Ângelo, Loures, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Clinical information will be shared with co-investigators
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available for the intire study, 4 years
Access Criteria: Only health professionals from Hospital Beatriz Ângelo, that make parte of the trial team will have acess